CLINICAL TRIAL: NCT00904436
Title: Evaluation of Breathing Pattern and Dyspnea in Subjects With Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Spungen, Ann - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Factorial | Masking: None
Other Study IDs: B2648C-1
Record Dates: First submitted 2009-05-14; First posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Dyspnea; Tetraplegia
Keywords: Tetraplegia; Breathing Patterns; Dyspnea
MeSH Terms: conditions — Dyspnea; Quadriplegia | interventions — Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Spinal Cord Injury: subjects who have cervical spinal cord injury and complaints of dyspnea
  Interventions: Drug: ipratropium (Atrovent)
- 2 (No Intervention): Controls

INTERVENTIONS:
Drug: ipratropium (Atrovent) — Bronchodilator Treatment: Subjects will inhale 1 unit dose vial of aerosolized ipratropium (500 mcg of ipratropium (Atrovent) mixed in 2.5 ml of saline).
  Arms: 1

SUMMARY:
Breathlessness is an extremely common and uncomfortable symptom that is reported in more than two-thirds of persons with tetraplegia. This disordered pulmonary function is due to respiratory muscle paralysis or to sympathetic denervation results in a restrictive impairment and airway hyperreactivity, respectively. These restrictive and obstructive dysfunctions have been associated with the symptom of breathlessness. However, mechanisms contributing to dyspnea in persons who have tetraplegia are not well understood. It has been demonstrated that persons with tetraplegia have an increased prevalence of breathlessness and may have an altered breathing pattern. The purpose of this study is to determine the breathing pattern at rest and measure the changes in breathing after a bronchodilator treatment (a medicine commonly used to treat asthma that relaxes and opens up airways). The determination of breathing pattern is done by measuring the movements in the chest wall while breathing. This design will elucidate differences in breathing patterns between those with tetraplegia and controls, as well as demonstrate the effect of bronchodilatation on motor drive and timing. Knowledge of the intraindividual variability and mean values of the components of the breathing pattern will improve our understanding of breathlessness in these individuals.

DETAILED DESCRIPTION:
The goal of this study is to evaluate mechanisms of dyspnea in tetraplegia. This goal will be accomplished by completing the following specific objectives:

1. To noninvasively assess dyspnea, motor drive, and respiratory timing during prolonged periods of resting breathing.
2. To determine if relationships exist between these breathing pattern components and dyspnea.
3. To determine if the relationships among respiratory timing, drive, and dyspnea are altered by a bronchodilator and over its duration of action.

These specific objectives will be used to test the hypotheses that:

1. During prolonged periods of resting breathing, respiratory timing will be altered and motor drive will be increased and less variable than in able-bodied controls.
2. There will be a positive association between motor drive and dyspnea.
3. Improving respiratory mechanics by bronchodilator administration will reduce drive, normalize timing and lessen dyspnea over the duration of action of the drug.

Completion of the proposed studies will expand our existing knowledge of ventilatory control in persons with tetraplegia and relate these changes to dyspnea, a common and distressing clinical problem in these individuals. These studies will also provide a better characterization of breathing patterns and their intrasubject variability in persons with tetraplegia. Currently, the only information regarding breathing patterns in tetraplegia are of limited duration (15-30 minutes). If this pilot study reveals significant relationships between motor drive, timing, and dyspnea, compiling "normative" data for breathing patterns from large numbers of individuals with tetraplegia may be useful in evaluating dyspnea in different clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have cervical spinal cord injury
2. Complaints of dyspnea
3. Healthy non-paralyzed controls

Exclusion Criteria:

1. Active pulmonary infection
2. Current history of chronic pulmonary disease or asthma
3. Current smoker (> 0.5 ppd)
4. Age < 18 or > 60 years
5. Duration of spinal cord injury < 1 year
6. Unable to sit upright in a chair or wheelchair for a full day
7. Persons taking anticholinergic (e.g., ditropan) or gaba (e.g., baclofen) agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1999-12; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
The goal of this study is to evaluate ventilatory control during quiet breathing in subjects with tetraplegia by obtaining dyspnea scores and noninvasively measuring indices of motor output (tidal volume / inspiratory time, VT/TI). | 2 years

SECONDARY OUTCOMES:
The goal of this study is to evaluate ventilatory control during quiet breathing in subjects with tetraplegia by obtaining dyspnea scores and noninvasively measuring indices of timing (inspiratory time/total breath time TI/TTOT). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Spungen, EdD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States